CLINICAL TRIAL: NCT07229846
Title: A Single-arm, Single-center, Phase II Clinical Study of Aipalolitovorelizumab (QL1706) Combined With Bevacizumab and Standard Chemotherapy as First-line Treatment for MSS/pMMR Metastatic Colorectal Cancer With BRAF V600E Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, professor, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-CRC-QIBA-3006
Record Dates: First submitted 2025-08-05; First posted 2025-11-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; BRAF V600E mutation; Microsatellite stability; Immunotherapy; First-line treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — XELOX; Bevacizumab; Oxaliplatin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm experimental group (Experimental)
  Interventions: Drug: Aipalolitovorelizumab; Drug: XELOX + Bevacizumab; Drug: mFOLFOX + Bevacizumab; Drug: FOLFOXIRI + Bevacizumab; Drug: Oxaliplatin + Irinotecan + Capecitabine + Bevacizumab

INTERVENTIONS:
Drug: Aipalolitovorelizumab — Aipalolitovorelizumab (QL1706) Injection: 5 mg/kg, intravenous infusion (ivgtt), d1, Q3W;
Drug: XELOX + Bevacizumab — Bevacizumab 7.5 mg/kg, intravenous infusion, Day 1; Oxaliplatin 130 mg/㎡, intravenous infusion over 2 hours, Day 1; Capecitabine 1000 mg/㎡, oral administration (po), twice a day (bid), Days 1-14. Repeat every 3 weeks.
Drug: mFOLFOX + Bevacizumab — Bevacizumab 5 mg/kg, intravenous infusion, Day 1; Oxaliplatin 85 mg/㎡, intravenous infusion over 2 hours, Day 1; Calcium Folinate 400 mg/m², intravenous infusion over 2 hours, Day 1; Fluorouracil 400 mg/m², intravenous bolus, Day 1, followed by 1200 mg/(m²·d) continuous intravenous infusion for 2 days (total dose 2400 mg/m², infusion over 46-48 hours). Repeat every 2 weeks.
Drug: FOLFOXIRI + Bevacizumab — Bevacizumab 5 mg/kg, intravenous infusion, Day 1; Irinotecan 165 mg/m², intravenous infusion, Day 1; Oxaliplatin 85 mg/m², intravenous infusion, Day 1; Calcium Folinate 400 mg/m², intravenous infusion, Day 1; Fluorouracil with a total dose of 2400-3200 mg/m², continuous intravenous infusion over 48 hours on Day 1. Repeat every 2 weeks.
Drug: Oxaliplatin + Irinotecan + Capecitabine + Bevacizumab — Bevacizumab 7.5 mg/kg, intravenous infusion, Day 1; Oxaliplatin 130 mg/㎡, intravenous infusion over 2 hours, Day 1; Irinotecan 180 mg/m², intravenous infusion over 30-90 minutes, Day 1; Capecitabine 1000 mg/㎡, oral administration (po), twice a day (bid), Days 1-14. Repeat every 3 weeks.

SUMMARY:
This is an open-label, single-arm, single-center phase II clinical study, aiming to investigate the safety and efficacy of Aipalolitovorelizumab (QL1706) combined with bevacizumab plus standard chemotherapy regimen as first-line treatment for patients with MSS/pMMR metastatic colorectal cancer harboring BRAF V600E mutation.

Patients will receive intravenous administration of Aipalolitovorelizumab (QL1706) injection + bevacizumab + oxaliplatin/irinotecan/fluorouracil/calcium folinate, along with oral capecitabine. After completing the corresponding treatment cycles, patients will enter the maintenance treatment phase as determined by the researcher. In the maintenance treatment phase, a 3-week treatment regimen of Aipalolitovorelizumab (QL1706) injection combined with bevacizumab and capecitabine will be adopted, with the administration method and dosage remaining unchanged.

The primary endpoint of this study is objective response rate (ORR); the secondary endpoints include progression-free survival (PFS), overall survival (OS), disease control rate (DCR), duration of response (DOR), and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (inclusive of 18 and 75 years) at the time of signing the ICF, male or female;
2. Patients with histopathologically confirmed unresectable metastatic colorectal adenocarcinoma of MSS/pMMR type with known BRAF V600E mutation;
3. Expected survival period ≥ 12 weeks;
4. No prior systemic antineoplastic drug treatment for metastatic colorectal adenocarcinoma (if the patient has previously received XELOX chemotherapy while waiting for genetic testing results, and meets other inclusion criteria as assessed by the researcher, they can be enrolled in the treatment);
5. For subjects who have received neoadjuvant/adjuvant therapy previously, the time from the last treatment to recurrence or progression must exceed 6 months;
6. Adverse events (AEs) related to previous treatment have recovered to grade ≤ 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) (except for alopecia);
7. According to the RECIST version 1.1 criteria, the researcher assesses that there is at least one measurable lesion, which should not have received local treatment such as radiotherapy (lesions located in the previously irradiated area can also be regarded as eligible measurable lesions if progression is confirmed);
8. Routine blood tests: No blood transfusion or use of blood products within 14 days. White blood cell count > 3000/µl, absolute neutrophil count (ANC) ≥ 1500 cells/µl, platelet count ≥ 75,000/µl, hemoglobin ≥ 9.0 g/dL, left ventricular ejection fraction (LVEF) ≥ 50%, Fridericia-corrected QT interval (QTcF) < 470 milliseconds, activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal (ULN);
9. Bilirubin ≤ 1.5 times ULN, ALT and AST ≤ 2.5 times ULN; if there is liver metastasis, ALT and AST ≤ 5 times ULN, total bilirubin (TBLL) ≤ 3 times ULN; creatinine < 1.5 times ULN;
10. ECOG PS score of 0-1 within 7 days before the first administration of the study drug;
11. Hepatitis B surface antigen (HBsAg) (-) and hepatitis B core antibody (HBcAb) (-), and no active hepatitis is clinically determined. If HBsAg (+) or HBcAb (+), then hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be < 1000 copies/mL or 200 IU/mL (if the lower limit of detection in the research unit is > 200 IU/mL, subjects with results below the lower limit of detection can be enrolled);
12. Hepatitis C virus (HCV) antibody (-); if HCV antibody (+), HCV-RNA test must be negative for enrollment. Subjects with co-infection of hepatitis B and hepatitis C must be excluded (HBsAg or HBcAb positive, and HCV antibody positive);
13. For female subjects of childbearing potential, the blood pregnancy test within 7 days before the first drug administration must be negative. Female subjects of childbearing potential and male subjects whose partners are women of childbearing age need to use at least one medically recognized contraceptive method (such as intrauterine device, contraceptives, or condoms) during the study treatment period and until at least 3 months after the last use of Aipalolitovorelizumab (QL1706) and bevacizumab, and at least 6 months after the last use of chemotherapy (whichever occurs later);
14. Provide a signed ICF and be willing to comply with all research procedures and rules specified in the protocol;
15. Have good compliance and be cooperative with follow-up.

Exclusion Criteria:

1. Have other active malignant tumors within 5 years before the first administration of the study drug. Patients with cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, and carcinoma in situ of the breast can be enrolled;
2. Have central nervous system (CNS) or leptomeningeal metastasis;
3. Have received radiotherapy within 6 months before the start of study treatment; except for palliative radiotherapy for bone lesions performed more than 14 days before the start of study treatment; radiotherapy covering more than 30% of the bone marrow area within 28 days before the first administration is not allowed;
4. Have previously received treatment with targeted drugs against EGFR or VEGF/vascular endothelial growth factor receptor (VEGFR) targets (including bevacizumab, cetuximab, panitumumab, aflibercept, regorafenib, or biosimilars of the above drugs, etc.);
5. Have previously received any T-cell co-stimulation or immune checkpoint inhibitor therapy, including but not limited to CTLA-4 inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other T-cell-targeted drugs;
6. Have a known history of severe allergy to any study drug analogs or study drug excipients;
7. Pleural effusion, pericardial effusion that cannot be controlled by appropriate intervention, or ascites that requires frequent drainage;
8. Have had cerebrovascular accident, myocardial infarction, unstable angina, or poorly controlled arrhythmia (including QTc interval ≥ 450 ms in males and ≥ 470 ms in females) within half a year (QTc interval is calculated by Fridericia formula);
9. Have New York Heart Association (NYHA) class III or IV cardiac insufficiency, or echocardiography shows left ventricular ejection fraction (LVEF) < 50%;
10. Have a history of immunodeficiency, including positive human immunodeficiency virus (HIV) antibody test, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation;
11. Have active pulmonary tuberculosis;
12. Patients with past or current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of pulmonary function, etc., which may interfere with the detection and treatment of suspected drug-related pulmonary toxicity;
13. Have active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes). Except for the following subjects: patients with vitiligo or cured childhood asthma/allergies who do not need any intervention in adulthood; patients with autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone; type I diabetes mellitus using a stable dose of insulin;
14. Have received live attenuated vaccine treatment within 28 days before the first administration of the study drug;
15. Subjects who need continuous systemic treatment (> 7 days) with corticosteroids (> 10 mg/day prednisone or equivalent dose of similar drugs) or other immunosuppressants within 14 days before the first administration of the study drug or during the study period. In the absence of active autoimmune diseases, inhalation or topical use of steroids, or adrenal hormone replacement with a dose ≤ 10 mg/day prednisone equivalent dose is allowed;
16. Have had a severe infection (CTCAE > grade 2) within 4 weeks before the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; baseline chest imaging suggests active pulmonary inflammation accompanied by clinically relevant symptoms or signs; have symptoms and signs of infection within 2 weeks before the first use of the study drug, or require oral or intravenous antibiotic treatment, except for the case of prophylactic use of antibiotics;
17. Have received major surgery within 28 days before the first administration of the study drug. Major surgery in this study is defined as surgery that requires at least 3 weeks of recovery before being able to receive treatment in this study;
18. Have previously received intestinal stent implantation, and the intestinal stent has not been removed by the screening period;
19. Have hypertension that cannot be controlled by clinical treatment (i.e., systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
20. Have a history of hypertensive crisis or hypertensive encephalopathy;
21. CT/MRI images show that the tumor surrounds or invades the lumen of large blood vessels (such as pulmonary artery or superior vena cava);
22. Patients with a significant/severe bleeding history within 1 month before screening, or who received blood transfusion within 2 weeks before screening;
23. Currently using or have used aspirin (> 325 mg/day) or dipyridamole, ticlopidine, clopidogrel, and cilostazol for treatment within 7 days before the first administration of the study drug;
24. Currently using or have used full-dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes within 7 days before the first administration of the study drug. Prophylactic anticoagulation for open intravenous infusion systems is allowed, as long as the drug activity results in an international normalized ratio (INR) < 1.5×upper limit of normal (ULN) and activated partial thromboplastin time (APTT) within the normal range within 14 days before the first administration of the study drug. Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is allowed;
25. Need long-term daily administration of non-steroidal anti-inflammatory drugs (NSAIDs). Occasional use of NSAIDs to relieve medical symptoms such as headache or fever is allowed;
26. Have evidence of intra-abdominal gas that cannot be explained by puncture or recent surgery;
27. Have severe, unhealed or dehisced wounds, active ulcers, or untreated fractures;
28. Have had the following diseases within 6 months before the first administration of the study drug:

    1. Abdominal or tracheoesophageal fistula, gastrointestinal perforation or intra-abdominal abscess, and a large amount of ascites as judged by the researcher (defined as patients requiring drainage or treatment within two weeks);
    2. Intestinal obstruction and/or have had clinical signs or symptoms of gastrointestinal obstruction, including incomplete obstruction related to the original disease or requiring regular parenteral hydration, parenteral nutrition, or tube feeding. Patients with a history of incomplete obstruction/obstruction syndrome/intestinal obstruction signs/symptoms who have improved after treatment can be enrolled as assessed by the researcher;
    3. Severe, uncontrollable intra-abdominal inflammation judged by the researcher to require clinical intervention;
    4. Major vascular diseases (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis);
29. Have a known history of psychiatric drug abuse or drug addiction;
30. Any other diseases, clinically significant metabolic abnormalities, abnormal physical examination or laboratory test results, which, in the researcher's judgment, reasonably suggest that the patient has a disease or condition unsuitable for the use of the study drug (such as having epileptic seizures requiring treatment), or will affect the interpretation of study results, or put the patient at high risk;
31. Currently participating in other clinical studies, or the time between the planned start of treatment in this study and the end of treatment with drugs in the previous clinical study is less than 14 days;
32. Any factors affecting oral administration;
33. Patients deemed inappropriate for inclusion in this study by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR) andpartial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Defined as the time between signing the informed consent form to the disease progression (according to REClST v1.1 criteria) or death due to any cause
Disease Control Rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR),. partiaresponse (PR), and stable disease (SD) according to RECIST V1.1.
Duration of Response | 6 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.
Overall survival | 2 years
  Defined as the time between signing the informed consent form to death due tovarious causes.
Safety | 6 months
  Use NCI-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hosptital, Harbin, China